CLINICAL TRIAL: NCT06703411
Title: Intravenous Iron Sucrose for Acute Decompensated Heart Failure Patients With Reduced Ejection Fraction and Iron Deficiency
Acronym: IronSucroseHF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cheng-Hsin General Hospital (Other)
Responsible Party: Principal Investigator, Hung-Yu Chang, Cardiologist, Cheng-Hsin General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHGH_IronSucrose_HFrEF_ID
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure With Reduced Ejection Fraction (HFrEF); Hospitalization; Iron Deficiency
Keywords: Heart failure; Iron sucrose; Hospitalization; Quality of life
MeSH Terms: conditions — Iron Deficiencies; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron sucrose (Experimental): IV iron sucrose 200mg per visit
  Interventions: Drug: Iron Sucrose IV; Drug: Standard Medical Therapy
- Standard of care (Active Comparator): Standard of care (HFrEF4 pillars treatment)
  Interventions: Drug: Standard Medical Therapy

INTERVENTIONS:
Drug: Iron Sucrose IV — IV iron sucrose 200mg per visit
  Arms: Iron sucrose
Drug: Standard Medical Therapy — Standard of care (HFrEF 4 pillars treatment)

SUMMARY:
Iron deficiency (ID) affects about 25% of the global population, presenting with symptoms of fatigue, weakness, and impaired cognitive function. Its prevalence is lower in developed regions, due to fortified foods, supplements, and better healthcare. In contrast, ID is more common in resource-limited countries, where diets lack iron, healthcare is less accessible, and infections like malaria and hookworm are more prevalent. In Asia, ID rates vary widely, influenced by dietary habits, socioeconomic factors, and healthcare quality.

The concurrent presence of ID and heart failure (HF) is increasingly acknowledged as a significant clinical issue, leading to a worsened prognosis and diminished quality of life for those affected. Recent research has reported a high prevalence of ID among HF patients, ranging from 30% to 50%, depending on the population studied and the diagnostic criteria used. Furthermore, ID in HF is linked with increased disease severity, higher hospitalization rates, and a greater risk of mortality. Interestingly, the prevalence of co-existing ID among HF patients does not vary between Western and Asian cohorts.

Recent clinical trials involving the supplement of ferric carboxymaltose have shown the effectiveness of intravenous iron therapy in enhancing exercise capacity, improving quality of life, and reducing HF-related hospitalizations in patients with heart failure and reduced ejection fraction (HFrEF) and ID. The European and American guidelines both recommend routine screening for ID in HFrEF patients and suggest considering iron carboxymaltose for those with ID to improve clinical outcomes.

Despite the importance of addressing ID in HF for optimizing patient care and improving prognosis, in many countries, due to the high price of iron carboxymaltose, only iron sucrose is available for intravenous iron supplementation, which is contrary to current guidelines. The efficacy and safety of intravenous iron sucrose in patients with HF and ID were demonstrated in the FERRIC-HF trial, but this study was conducted more than a decade ago. In an era marked by significant changes in HF treatment approaches, it remains unclear whether intravenous iron sucrose provides benefits to HF patients receiving current treatment. In this study, our objective is to examine the impact of intravenous iron sucrose on acutely decompensated HFrEF patients with co-existing ID, with a focus on improvements in iron profiles and quality of life. Our hypothesis suggests that, despite advancements in standard HF treatments, the additional use of intravenous iron sucrose could lead to an improved quality of life among HFrEF patients with ID.

ELIGIBILITY:
Inclusion criteria were: (1) adult patients admitted with acute decompensated HFrEF (i.e., a left ventricular ejection fraction [LVEF] of less than 40%) and New York Heart Association (NYHA) functional class II or III symptoms; and (2) patients meeting the laboratory criteria for ID at hospitalization, defined as ferritin levels below 100 ng/mL, or ferritin levels between 100 and 299 ng/mL with transferrin saturation (TSAT) below 20%.

- Exclusion criteria included: (1) hemoglobin levels of 15 g/dL or higher; (2) refusal to participate; (3) active infection or bleeding; (4) concomitant oral iron treatment; and (5) terminal illness with an expected lifespan under 6 months.

-

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
KCCQ score (quality of life) | 4 weeks
  KCCQ score (quality of life)

SECONDARY OUTCOMES:
Iron profiles | 4 weeks
  Iron profiles, including ferritin, iron, TIBC, TSAT

CONTACTS AND LOCATIONS:
Locations (1):
- Cheng Hsin General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ponikowski P, Anker SD, AlHabib KF, Cowie MR, Force TL, Hu S, Jaarsma T, Krum H, Rastogi V, Rohde LE, Samal UC, Shimokawa H, Budi Siswanto B, Sliwa K, Filippatos G. Heart failure: preventing disease and death worldwide. ESC Heart Fail. 2014 Sep;1(1):4-25. doi: 10.1002/ehf2.12005. PMID 28834669
- [Derived] Sung HP, Yin WH, Chen SF, Hung CL, Lin KC, Chang HY. Intravenous Iron Sucrose for Acute Decompensated Heart Failure Patients with Reduced Ejection Fraction and Iron Deficiency. Rev Cardiovasc Med. 2025 Apr 17;26(4):28216. doi: 10.31083/RCM28216. eCollection 2025 Apr. PMID 40351678